CLINICAL TRIAL: NCT01643941
Title: A Phase 1/2 Placebo-controlled, Randomized, Double-blind Trial To Evaluate The Safety, Tolerability, And Immunogenicity Of 3 Ascending Dose Levels Of A 4-antigen Staphylococcus Aureus Vaccine (sa4ag) And A Single Dose Level Of A 3-antigen Staphylococcus Aureus Vaccine (sa3ag) In Healthy Adults Aged 65 To <86 Years
Brief Title: Evaluation of a Single Vaccination of One of Three Ascending Dose Levels of a 4-Antigen Staphylococcus Aureus Vaccine (SA4Ag) and a Single Dose Level of a 3-Antigen Staphylococcus Aureus Vaccine (SA3Ag) in Healthy Adults Aged 65 to <86 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: B3451011
Record Dates: First submitted 2012-07-09; First posted 2012-07-18 (Estimated); Last update posted 2019-03-04 (Actual); Status verified 2019-02

CONDITIONS: Staphylococcal Infections
Keywords: Staphylococcus aureus; vaccine; Staphylococcal infection
MeSH Terms: conditions — Staphylococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental): SA4Ag vaccine low dose
  Interventions: Biological: SA4Ag vaccine low dose; Procedure: Blood draw; Procedure: Colonization swab sample
- 2 (Experimental): SA4Ag vaccine mid dose
  Interventions: Biological: SA4Ag vaccine mid dose; Procedure: Blood draw; Procedure: Colonization swab sample
- 3 (Experimental): SA4Ag vaccine high dose
  Interventions: Biological: SA4Ag vaccine high dose; Procedure: Blood draw; Procedure: Colonization swab sample
- 4 (Experimental): SA3Ag vaccine
  Interventions: Biological: SA3Ag vaccine; Procedure: Blood sample; Procedure: Colonization swab sample
- 5 (Placebo Comparator): Placebo
  Interventions: Biological: Placebo; Procedure: Blood draw; Procedure: Colonization swab samples

INTERVENTIONS:
Biological: SA4Ag vaccine low dose — Subjects receive 1 intramuscular injection (0.5 mL) of the low dose level of the SA4Ag vaccine.
  Arms: 1
Procedure: Blood draw — Blood for HIV, HBV and HCV screening will be collected prior to enrollment for Phase 1 subjects. Blood for hematology, coagulation and blood chemistry will be collected at a minimum of 3 timepoints from Phase 1 subjects. Blood for immunogenicity will be collected from all subjects at various timepoints.
  Arms: 1
Procedure: Colonization swab sample — Colonization swabs will be collected from all subjects at various timepoints.
  Arms: 1
Biological: SA4Ag vaccine mid dose — Subjects receive 1 intramuscular injection (0.5 mL) of the mid dose level of the SA4Ag vaccine.
  Arms: 2
Procedure: Blood draw — Blood for HIV, HBV and HCV screening will be collected prior to enrollment for Phase 1 subjects. Blood for hematology, coagulation and blood chemistry will be collected at a minimum of 3 timepoints from Phase 1 subjects. Blood for immunogenicity will be collected from all subjects at various timepoints.
  Arms: 2
Procedure: Colonization swab sample — Colonization swabs will be collected from all subjects at various timepoints.
  Arms: 2
Biological: SA4Ag vaccine high dose — Subjects receive 1 intramuscular injection (0.5 mL) of the high dose level of the SA4Ag vaccine.
  Arms: 3
Procedure: Blood draw — Blood for HIV, HBV and HCV screening will be collected prior to enrollment for Phase 1 subjects. Blood for hematology, coagulation and blood chemistry will be collected at a minimum of 3 timepoints from Phase 1 subjects. Blood for immunogenicity will be collected from all subjects at various timepoints.
  Arms: 3
Procedure: Colonization swab sample — Colonization swabs will be collected from all subjects at various timepoints.
  Arms: 3
Biological: SA3Ag vaccine — Phase 2 only: Subjects receive 1 intramuscular injection (0.5 mL) of the mid dose level of the SA3Ag vaccine.
  Arms: 4
Procedure: Blood sample — Blood for immunogenicity will be collected from all subjects at various timepoints.
  Arms: 4
Procedure: Colonization swab sample — Colonization swabs will be collected from all subjects at various timepoints.
  Arms: 4
Biological: Placebo — Subjects receive one intramuscular injection (0.5 mL) of placebo which contains excipients of the vaccine formulation minus the active ingredients.
  Arms: 5
Procedure: Blood draw — Blood for HIV, HBV and HCV screening will be collected prior to enrollment for Phase 1 subjects. Blood for hematology, coagulation and blood chemistry will be collected at a minimum of 3 timepoints from Phase 1 subjects. Blood for immunogenicity will be collected from all subjects at various timepoints.
  Arms: 5
Procedure: Colonization swab samples — Colonization swabs will be collected from all subjects at various timepoints.
  Arms: 5

SUMMARY:
This is a Phase 1 and Phase 2 study of a single vaccination with one of three dose levels of a 4-antigen investigational vaccine against Staphylococcus aureus (SA4Ag) and a single dose level of a 3-antigen Staphylococcus aureus vaccine (SA3Ag). The main goal of the study is to determine how safe and well tolerated the vaccine is as well as to describe the immune response elicited by the vaccine in healthy adults aged 65 to <86 years. In addition, the study aims to assess the effect of the Staphylococcus aureus vaccine on the presence of the Staphylococcus aureus within the nose, throat and perineal skin of healthy adults aged 65 to <86 years.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males and healthy postmenopausal females, aged 65 to <86 years at enrollment, as determined by medical history, physical examination, and the clinical judgment of the investigator to be eligible for the study. Subjects with preexisting chronic medical conditions determined to be stable may be included.
* Available for the entire duration of the study, and able to comply with scheduled visits, study plan, laboratory tests, and other study procedures including completion of the electronic diary (e diary) from Day 1 to Day 14 following vaccination.
* Able to be contacted by telephone during study participation.
* Male subjects who, in the opinion of the investigator, are biologically capable of fathering children, and who are sexually active with women of childbearing potential must agree to use a highly effective method of contraception throughout the study.

Exclusion Criteria:

* Unstable chronic medical condition or disease requiring significant change in therapy or hospitalization for worsening disease within 3 months before receipt of study vaccine.
* Serious chronic medical disorders or any disorder that in the investigator's opinion precludes the subject from participating in the study.
* Donation of blood volume of 250 mL or greater or donation of plasma within 3 months prior to enrollment through conclusion of the study.
* Bleeding condition associated with prolonged bleeding time that may contraindicate intramuscular injection or blood draw including subjects taking anticoagulant, antiplatelet and/or antithrombotic agents except for low-dose daily aspirin within 30 days before enrollment through completion of Visit 6 (Day 29).
* Any contraindication to vaccination or vaccine components, including previous anaphylactic reaction to any vaccine or vaccine related components.
* Immunocompromised persons or subjects currently on immunosuppressive therapy or with a history of immunosuppressive therapy. History of immune-modifying drugs.
* Previous administration of S. aureus vaccination.
* Any infection proven or suspected to be caused by S. aureus within 6 months preceding study vaccination.
* Receipt of blood products or immunoglobulins (including monoclonal antibodies) within 12 months before enrollment through conclusion of the study.
* Participation in other investigational or interventional studies within 30 days before the current study begins and/or during study participation. Participation in purely observational studies is acceptable.
* Subjects who are investigational site staff members or subjects who are immediate family members (first-degree relatives) of investigational site staff members or Pfizer employees directly involved in the conduct of the trial.
* Residence in a nursing home or long-term care facility or requirement for semiskilled nursing care. An ambulatory subject who is a resident of a retirement home or village is eligible for the trial.
* A Mini-Mental State Examination (MMSE) score of ≤21.
* For Phase 1 subjects only, any abnormality in screening hematology, coagulation, and/or blood chemistry laboratory values except as noted in protocol
* Subjects with known active disease with human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV), or Phase 1 subjects with a positive screening test for HIV, HBV and/or HCV.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Planned surgical procedure within 30 days following vaccination.

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 284 (Actual)
Dates: Start 2012-08; Primary Completion 2013-05 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Number and proportion of subjects reporting solicited local reactions (size of redness and/or swelling and severity of pain at the injection site) and severity of the local reactions as self-reported on electronic diaries (e-diaries) | 14 days
Number and proportion of subjects reporting solicited systemic events (fever, vomiting, diarrhea, headache, fatigue, new or worsening muscle pain, new or worsening joint pain) and severity of solicited systemic events self-reported on electronic diaries | 14 days
Number and proportion of subjects reporting unsolicited AEs and serious adverse events (SAEs) categorized according to the Medical Dictionary for Regulatory Activities (MedDRA) | 1 month (AEs); 6 months (SAEs)
Number and proportion of Phase 1 subjects with abnormal hematology, coagulation and blood chemistry lab assessments | 14 days
Number and proportion of Phase 1 subjects with grading shifts in hematology, coagulation and blood chemistry laboratory assessments | 14 days
Proportion of subjects achieving antibody responses to specific vaccine components with results ≥ thresholds defined for each vaccine component based on immunoglobulin-binding and/or opsonphagocytic activity assays | 1 month

SECONDARY OUTCOMES:
Immunoglobulin titers measured as geometric mean titers for each antigen at each applicable blood sampling time point, as measured by antigen-specific antibody levels using an immunoglobulin binding assay. | various, up to 12 months
Opsonophagocytic activity titers measured as geometric mean titers against S. aureus isolates at each applicable blood sampling time point. | various, up to 12 months
Immunoglobulin geometric mean fold rise for each of the vaccine components as measured by antigen-specific antibody levels using an immunoglobulin binding assay. | 1 month
Geometric mean fold rise on opsonophagocytic activity assay titers against S. aureus isolates. | 1 month
Proportion of subjects achieving antibody responses to specific antigens with results ≥ thresholds defined for each vaccine component at each applicable visit. | Various, up to 12 months
Proportion of subjects with ≥2-fold, ≥4-fold, ≥8-fold, ≥16-fold, and ≥32-fold increase in immunoglobulin titers from baseline to each applicable visit after vaccination for each antigen. | Various, up to 12 months
Proportion of subjects with ≥2-fold, ≥4-fold, ≥8-fold, ≥16-fold, and ≥32-fold increase in opsonophagocytic activity titers against S. aureus isolates from baseline to each applicable visit after vaccination. | Various, up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (7):
- United States (7):
  - Broward Research Group, Hollywood, Florida
  - Miami Research Associates, South Miami, Florida
  - Vince and Associates Clinical Research, Overland Park, Kansas
  - PMG Research of Raleigh, LLC, Cary, North Carolina
  - Cincinnati Children's Hospital Medical Center Gamble Program for Clinical Studies, Cincinnati, Ohio
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Benchmark Research, Austin, Texas

REFERENCES:
- [Derived] Creech CB, Frenck RW, Fiquet A, Feldman R, Kankam MK, Pathirana S, Baber J, Radley D, Cooper D, Eiden J, Gruber WC, Jansen KU, Anderson AS, Gurtman A. Persistence of Immune Responses Through 36 Months in Healthy Adults After Vaccination With a Novel Staphylococcus aureus 4-Antigen Vaccine (SA4Ag). Open Forum Infect Dis. 2019 Dec 24;7(1):ofz532. doi: 10.1093/ofid/ofz532. eCollection 2020 Jan. PMID 31993453
- [Derived] Creech CB, Frenck RW Jr, Sheldon EA, Seiden DJ, Kankam MK, Zito ET, Girgenti D, Severs JM, Immermann FW, McNeil LK, Cooper D, Jansen KU, Gruber W, Eiden J, Anderson AS, Baber J. Safety, tolerability, and immunogenicity of a single dose 4-antigen or 3-antigen Staphylococcus aureus vaccine in healthy older adults: Results of a randomised trial. Vaccine. 2017 Jan 5;35(2):385-394. doi: 10.1016/j.vaccine.2016.11.032. Epub 2016 Nov 17. PMID 27866765
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B3451011&StudyName=Evaluation%20of%20a%20Single%20Vaccination%20of%20One%20of%20Three%20Ascending%20Dose%20Levels%20of%20a%204-Antigen%20Staphylococcus%20aureus%20Vaccine%20%28SA4Ag%29%20and%20